CLINICAL TRIAL: NCT01063400
Title: OS09328 Feasibility Study: Comparison of Performance Status With Objective Physical Activity Monitors
Brief Title: Feasibility Study: Comparison of Performance Status With Objective Physical Activity Monitors
Status: Terminated | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: OS09328
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Activity monitoring
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — monitoring of physical activity for 14 days using physical activity monitoring devices along with activity diary

SUMMARY:
The purpose of this research is to examine the relationship between performance status rating and the actual amount of physical activity a subject does when it is measured by an activity monitor.

ELIGIBILITY:
Inclusion Criteria:

* Worst Daily Pain rating of < 4/10
* ECOG Performance Status of 0, 1, or 2
* Prior malignancy is allowed as long as it is inactive or well-controlled without current anti-tumor therapy required

Exclusion Criteria:

* Known brain metastasis
* Use of assistive devices (cane, crutch)
* No concurrent radiotherapy: all radiotherapy must be completed 4 weeks prior to enrollment in this study
* Patients receiving only targeted therapy are not eligible(e.g.erlotinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients receiving chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of examining physical activity (through objective measurement devices) and performance status in a 14-day study of lung cancer patients. | 14 days

SECONDARY OUTCOMES:
To determine the number of days of monitoring necessary to reliably estimate energy expenditure (steps/day, and % of time spent sedentary) in lung cancer patients undergoing chemotherapy. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Toby Campbell, MD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States